CLINICAL TRIAL: NCT06769009
Title: The Next Step Towards the Elimination of Iodine Deficiency and Preventable Iodine-related Disorders in Europe
Brief Title: EUthyroid2: the Next Step Towards the Elimination of Iodine Deficiency and Preventable Iodine-related Disorders in Europe
Acronym: EUthyroid2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EUthyroid (Other)
Collaborators: EU Horizon (Unknown); UK Research and Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 101095643
Record Dates: First submitted 2024-11-21; First posted 2025-01-10 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Iodine Deficiency
Keywords: prevention; iodine deficiency; intervention study; cluster-randomized controlled trial; complex intervention; adaption to context; awareness; urinary iodine status; iodine intake; nutrition; education

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Educational intervention measures on iodine, iodine deficiency and iodine intake
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Educational intervention measures on iodine, iodine deficiency and iodine intake — The intervention consist of an educational intervention which will educate the young women on the importance of iodine, the consequences of iodine deficiency, dietary iodine sources and the iodine in pregnancy. The educational intervention consist of four intervention components: an iodine feedback tool, and educational iodine conversation with a healthcare professional, an iodine factsheet and an iodine video. The healthcare professionals who carry out the educational conversation will receive a specially designed training program.
  Arms: Intervention Group

SUMMARY:
In EUthyroid2 intervention measures are to be developed, implemented in ambulatory care settings and evaluated to effectively raise awareness for the risks of iodine deficiency among young women (18-24 years) in three European countries (Norway, Poland, UK) as well as Bangladesh and Pakistan. A cluster-randomized controlled trial with three points of measurements will be applied in each participating country. The intervention will be adapted to the different contextual characteristics of the implementation sites. A process evaluation with a convergent parallel mixed methods design will be conducted. For this, participants and healthcare professionals will be surveyed and semi-structured interviews will be carried out.

DETAILED DESCRIPTION:
BACKGROUND: Iodine deficiency (ID) is a leading risk factor for the development of thyroid disorders, of which in particular women are affected. During pregnancy, ID can increase the risk of developmental disorders in the offspring, however, it is considered as one of the most preventable causes of mental impairment in children. Therefore, the EUthyroid2 project aims to contribute to the prevention of ID and associated symptom and disease burden in adolescence and young women in Europe and beyond.

AIM: An educational intervention is to be developed, implemented in ambulatory care settings and evaluated to effectively raise awareness for the risks of ID among young women (18-24 years) in three European countries (Norway, Poland, UK) as well as Bangladesh and Pakistan.

METHODS: A cluster-randomised controlled trial is to be conducted in each of the five countries. 10 clusters per country (5 intervention group clusters and 5 control group clusters) are planned to achieve a final sample size of 200 study participants per implementing country with one baseline (before the intervention) and two follow-up measurements (2-4 weeks and 6-8 months after the intervention). In all, 1000 participants are to be recruited and data for all measurement points collected. Due to differences in the healthcare systems, the ambulatory care units, where the intervention will be implemented, may vary across the countries. Before recruiting the women, the healthcare professionals who carry out the intervention will receive a specially designed training program. To assure the intervention's functionality and effectiveness, recommendations for the development of complex interventions, appropriate theories and frameworks will be considered and a context analysis will be conducted. The primary outcome of the study is iodine awareness and knowledge measured by a newly developed questionnaire. Other outcomes includes measurement of iodine status (urinary iodine concentration), intake of dietary iodine sources (measured by a food frequency questionnaire), and iodine related behaviours. Sociodemographic characteristics and general dietary habits will also be measured. Descriptive analyses for all variables will be performed. Intervention groups will be compared to control groups over time to test effectiveness. Subgroup and country-specific analyses will also be computed. A process evaluation will be conducted to evaluate the implementation process with a convergent parallel mixed methods design. For this, healthcare professionals in the ambulatory care settings and the women who received the intervention will be invited to participate in an online survey. Further, ca. 20-30 semi-structured interviews will be conducted with women and healthcare professionals.

CONCLUSION / OUTLOOK: The project results may support health authorities across countries to implement effective measures to reduce ID and associated risks. This may sustainably reduce the disease burden induced by ID for young women, pregnant women and their offspring.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant Female
* Age 18-24 years at the time point of recruitment
* Attending the specified settings
* Sufficient language skills to understand the study information, informed consent and the questionnaire

Exclusion Criteria:

* Having a thyroid disease
* Pregnancy at the timepoint of recruitment and during the intervention period
* Lactation

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Significant change in awareness of iodine in women (18-24 years) within the intervention group from T1 (baseline) to T2 (2-4 weeks) and T3 (6-8 months) and compared to women (18-24 years) in the control group. | T1 = baseline (before the intervention); T2 = first follow-up (2-4 weeks after the intervention); T3 = second follow-up (6-8 months after the intervention)
  Difference in iodine awareness is measured by an iodine awareness questionnaire. The scoring ranges from 1 to 22 points with higher scores indicating a better outcome of awareness.
  The difference in iodine awareness in women (18-24 years) is examined:
  1. within the intervention group from:
     * T1 (baseline) compared to T2 (2-4 weeks after the intervention)
     * T1 (baseline) compared to T3 (6-8 months after the intervention)
  2. in the intervention compared to the control group at:
     * T2 (2-4 weeks after the intervention)
     * T3 (6-8 months after the intervention)

SECONDARY OUTCOMES:
Significant change in the urinary iodine status of women (18-24 years) within the intervention group from T1 (baseline) to T2 (2-4 weeks) or T3 (6-8 months) and compared to women (18-24 years) in the control group | T1 = baseline (before the intervention); T2 = first follow-up (2-4 weeks after the intervention); T3 = second follow-up (6-8 months after the intervention)
  The urinary iodine concentration will be measured on a scale from 0- to n (there is no maximum value). The median UIC will be compared against the WHO classification of adequate iodine intake of a median UIC ≥100 µg/L and will be compared within the interention group and at each time-point between the intervention and control group.
  Difference in iodine status (measured by UIC in µg/L) of women (18-14 years) is examined:
  1. within the intervention group before and after the intervention:
     * T1 (baseline) compared to T2 (2-4 weeks after the intervention)
     * T1 (baseline) compared to T3 (6-8 months after the intervention)
  2. in the intervention group compared to the control group at:
     * T2 (2-4 weeks after the intervention)
     * T3 (6-8 months after the intervention)
Significant change in intake of dietary iodine sources of women (18-24 years) within the intervention group from T1 (baseline) to T2 (2-4 weeks) or T3 (6-8 months) and compared to women (18-24 years) in the control group | T1 = baseline (before the intervention); T2 = first follow-up (2-4 weeks after the intervention); T3 = second follow-up (6-8 months after the intervention)
  Differences in intake of dietary iodine sources is measured by a food frequency questionnaire (FFQ).Dietary iodine intake is assessed through a food frequency questionnaire (FFQ), covering five main categories (cow's milk, fish, eggs, supplements, and salt) and regional components in each country. Each category is scored based on frequency (portions per day, week, or month), and individual sources are analyzed for iodine intake.
  Difference in the FFQ of women (18-24 years) is examined:
  1. within the intervention group before and after the intervention:
     * T1 (baseline) compared to T2 (2-4 weeks after the intervention)
     * T1 (baseline) compared to T3 (6-8 months after the intervention)
  2. in the intervention group compared to the control group at:
     * T2 (2-4 weeks after the intervention)
     * T3 (6-8 months after the intervention)
  The outcomes will be analyzed statistically based on the different answers in the questionnaire and regional differences.
Significant change in awareness of iodine of healthcare professionals before (T1) and after the training (T2) | T1 = baseline (before the training); T2 = follow-up (2-4 weeks after the training)
  Difference in iodine awareness is measured by an iodine awareness questionnaire. The scoring ranges from 1 to 22 points with higher scores indicating a better outcome of awareness.
  Difference in iodine awareness of the healthcare professional is examined before and after the training:
  - T1 (baseline) compared to T2 (2-4 weeks after the intervention)
Significant change in intake of dietary iodine sources of the healthcare professional before (T1) and after the training (T2) | T1 = baseline (before the training); T2 = follow-up (2-4 weeks after the training)
  Dietary iodine intake is assessed through a food frequency questionnaire (FFQ), covering five main categories (cow's milk, fish, eggs, supplements, and salt) and regional components in each country. Each category is scored based on frequency (portions per day, week, or month), and individual sources are analyzed for iodine intake.
  Difference in the FFQ of healthcare professional is compared before and after the training:
  - T1 (baseline) compared to T2 (2-4 weeks after the intervention)

CONTACTS AND LOCATIONS:
Locations (6):
- Bangladesh University of Health, Dhaka, Bangladesh
- Institute of Marine Research, Bergen, Bergen, Norway
- Islamia College Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan
- Jagiellonian University, Krakow, Poland
- United Kingdom (2):
  - The Queen's University of Belfast, Belfast
  - University of Surrey, Guildford